CLINICAL TRIAL: NCT02579551
Title: Long Term Prospective Study Evaluating Effectiveness of Narrow Margins for Low-Risk Facial Basal Cell Carcinomas
Brief Title: Effectiveness of Narrow Margins in Patients With Low-Risk Basal Cell Carcinoma Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11D.479; NCI-2015-01624 (Registry Identifier: NCI Trial Identification); JT 2143 (Other: JeffTrial Number)
Record Dates: First submitted 2015-10-12; First posted 2015-10-19 (Estimated); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Skin Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (surgical excision) (Experimental): Patients undergo surgical excision of the skin lesion consisting of 1 and 2 mm circumferential margins during visit 1.
  Interventions: Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Procedure: Therapeutic Conventional Surgery — Undergo surgical excision

SUMMARY:
This clinical trial studies the effectiveness of narrow margins in patients with low-risk basal cell carcinoma undergoing surgery to remove skin lesions on the face. A margin is the area of normal tissue around a tumor taken out during surgery to make sure all of the cancer is removed. This clinical trial studies tissue samples to determine the least amount of tissue that must be removed to give an acceptable cure rate. This may allow less normal tissue to be removed from patients and may be a less expensive surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the success rate of narrow margin excisions of low-risk facial basal cell carcinoma (BCC).

SECONDARY OBJECTIVES:

I. To determine the narrowest excision margin for low-risk facial BCC that gives an acceptable (95%) cure rate over a 3 year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Location

   1. Area M (cheeks, forehead, scalp & neck) tumor size < 10 mm
   2. Area H (central face, eyelids, eyebrows, periorbital, nose, lips, chin, mandible, preauricular & postauricular, temple & ear) tumor size < 6 mm
2. Well-defined borders
3. Primary BCC
4. Patient is not immunosuppressed
5. There has not been prior radiotherapy to the site
6. Nodular subtype
7. No perineural involvement-(no neurological deficits grossly) -

Exclusion Criteria:

1. Location

   1. Area M tumor size > or = to 10 mm
   2. Area H tumor size > or = to 6 mm
2. Poorly defined borders
3. Recurrent BCC
4. Patient is immunosuppressed
5. There has been prior radiotherapy to the site -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2011-12-07 (Actual); Primary Completion 2014-02-01 (Actual); Study Completion 2017-05-04 (Actual)

PRIMARY OUTCOMES:
Success rate for 1 mm margins | Up to 3 years
  The success rate for 1 mm margin will be calculated along with an exact one-sided 95% confidence interval for the proportion. The success rate will be compared to a null value of 90% using a one-sided exact test of binomial proportion.
Success rate for 2 mm margins | Up to 3 years
  The success rate for 2 mm margin will be calculated along with an exact one-sided 95% confidence interval for the proportion. The success rate will be compared to a null value of 90% using a one-sided exact test of binomial proportion.

SECONDARY OUTCOMES:
Recurrence rate after 3 years | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lee, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson Univeristy, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/